CLINICAL TRIAL: NCT03016143
Title: A Randomized, Blinded, Comparative Study of Phase II Allantoic Split Inactivated Seasonal Influenza Vaccine in Healthy Adults
Brief Title: Immunogenicity and Safety Study of Allantoic Split Inactivated Seasonal Influenza Vaccine (VSI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: Asfendiyarov Kazakh National Medical University (Other); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VSI-II-01/2016
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2017-01

CONDITIONS: Influenza
Keywords: phase II; split; vaccine
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group #1 (Allantoic Split Inactivated Seasonal flu Vaccine) (Active Comparator): 100 volunteers aged 18 to 60 years, which introduced the vaccine allantoic split inactivated seasonal influenza
  Interventions: Biological: Allantoic Split Inactivated Seasonal flu Vaccine
- Group #2 (Allantoic Split Inactivated Seasonal flu Vaccine) (Active Comparator): 100 volunteers over the age of 60 years, which introduced the vaccine allantoic split inactivated seasonal influenza
  Interventions: Biological: Allantoic Split Inactivated Seasonal flu Vaccine
- Group #3 (Vaccine VAXIGRIP) (Experimental): 50 volunteers aged 18 to 60 years, which introduced vaccine VAXIGRIP
  Interventions: Biological: VAXIGRIP
- Group #4 (Vaccine VAXIGRIP) (Experimental): 50 volunteers over the age of 60 years, which introduced vaccine VAXIGRIP
  Interventions: Biological: VAXIGRIP

INTERVENTIONS:
Biological: Allantoic Split Inactivated Seasonal flu Vaccine — Allantoic split inactivated seasonal influenza vaccine has been prepared on eggs and is made from inactivated parts of the following influenza virus strains: NIBRG-121xp (A/California/7/2009 (H1N1)v and А/PR/8/34 (H1N1)), NYMC X-217 (A/ Victoria/361/2011(H3N2) and А/PR/8/34 (H1N1)), NYMC BX-49 (B/Texas/06/2011 (Yamagata lineage) - like High Yield Reassortant (1:1:6) With B/Lee/40 NP, B/Panama/45/90 NS genes).
  Arms: Group #1 (Allantoic Split Inactivated Seasonal flu Vaccine); Group #2 (Allantoic Split Inactivated Seasonal flu Vaccine)
Biological: VAXIGRIP — Vaxigrip - Seasonal Influenza, split virion, inactivated vaccine. Sanofi Pasteur Serial Number N3E681V
  Arms: Group #3 (Vaccine VAXIGRIP); Group #4 (Vaccine VAXIGRIP)

SUMMARY:
The study is a single centre, phase II, double-blind, randomized, comparative trial that explored the immunogenicity and safety of single dose a allantoic split inactivated seasonal influenza vaccine and VAXIGRIP vacccine in healthy adults the two age groups (in persons 18 to 60 years of age and older than 60 years).

ELIGIBILITY:
Inclusion Criteria:

* volunteers (men and women) aged 18 years and older.
* Literate and willing to provide written informed consent.
* A signed informed consent.

Exclusion Criteria:

* Available in anamnaze volunteer at any allergic reactions.
* Allergic reactions to chicken proteins, or any preceding vaccination.
* Acute illness with a fever (37.0 C).
* Vaccination against influenza in the 2015/2016 season.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Hypersensitivity after previous administration of any vaccine.
* History of chronic alcohol abuse and/or illegal drug use.
* Any clinically significant abnormal laboratory finding.
* A positive pregnancy test for all women of childbearing potential.
* Administration of immunosuppressive drugs or other immune modifying drugs within 4 weeks prior to study enrollment.
* Acute or chronic clinically significant pulmonary disease, cardiovascular disease, gastrointestinal disease, liver disease, neurological illness, liver disease, blood disease, skin disorder, endocrine disorder, neurological illness and psychiatric disorder as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of leukemia or any other blood or solid organ cancer.
* Receipt of antivirals, antibiotics, immunoglobulins or other blood products within 4 weeks prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Participation in another clinical trial within the previous three months or planned enrollment in such a trial during the period of this study.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Fold Increase in HI Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Geometric mean fold increase in HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination, as compared with Baseline.
Seroconversion Rate of Hemagglutination Inhibition (HI) Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Seroconversion rate was measured by hemagglutination inhibition (HI) antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Seroconversion rate was defined as the percentage of participants achieving a minimal 4-fold increase from the Baseline HI antibody titer in participants with a Baseline titer ≥10, or achieving an HI antibody titer of ≥40 in participants with a Baseline titer <10.
Seroprotection Rate of HI Antibody Titer | Change from Baseline HI Antibody Titer at 21 days
  Seroprotection rate, defined as the percentage of participants with HI antibody titer of ≥40, was measured by HI antibody titer for each of the three strains (A/H1N1 strain, A/H3N2 strain, B strain), 21 days after vaccination. Day 1 data is reported for reference.

SECONDARY OUTCOMES:
Percentage of Participants With Solicited Local and Systemic Adverse Events (AEs) | 21 Days
  Participants recorded solicited injection site and systemic adverse events in a Subject Diary. Solicited Locals AEs were: Injection Site Pain, Injection Site Redness, Injection Site Swelling, Injection Site Induration and Injection Site Ecchymosis. Solicited Systemic AEs were: Pyrexia, Malaise, Chills, Fatigue, Headache, Sweaty, Myalgia, Arthralgia, Nausea and Vomiting.
Percentage of Participants Reporting One or More Treatment-emergent Adverse Events (TEAE) | 21 Days
  Adverse events are defined as unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product, regardless of relationship to the medicinal product. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Percentage of Participants With Abnormal Safety Laboratory Tests at Least Once Post Dose Reported as AEs | 21 Days
  The percentage of participants with any abnormal standard safety laboratory values (Chemistry, Hematology and Urinalysis) collected throughout the study reported as AEs.
Serious adverse events (SAEs), including abnormal laboratory findings | 21 Days
  Serious adverse events (SAEs) are medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.

CONTACTS AND LOCATIONS:
Overall Officials: Berik M Khairullin, PhD, Principal Investigator — Research Institute for Biological Safety Problems
Locations (1):
- Kazakh National Medical University, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sarsenbayeva G, Issagulov T, Kassenov M, Abitay R, Orynbayev M, Stukova M, Pisareva M, Davlyatshin T, Lespek K, Khairullin B. Safety and immunogenicity of trivalent inactivated influenza vaccine in adults 60 years of age and older: a phase II, a randomized, comparative trial in Kazakhstan. Hum Vaccin Immunother. 2020 Aug 2;16(8):1791-1797. doi: 10.1080/21645515.2019.1705691. Epub 2020 Feb 12. PMID 32048890